CLINICAL TRIAL: NCT07158515
Title: The Heart Health After Cardiac Treatment Study
Acronym: HEART-ACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: This work was made possible by residual class settlement funds in the matter of April Krueger v. Wyeth, Inc., Case No. 03-cv-2496 (US District Court, SD of CA) (Unknown)
Responsible Party: Principal Investigator, Alexis Beatty, MD, Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-40216
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Rehabilitation
Keywords: comparative effectiveness; safety net

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored cardiac rehabilitation in a safety net setting (Experimental): A 12-week program of exercise training and health behavior counseling consisting of every other week group sessions (exercise and health behavior education) and every other week individual counseling sessions that address the cardiac rehabilitation core components.
  Interventions: Behavioral: Tailored cardiac rehabilitation
- Referral to an outside cardiac rehabilitation program (Active Comparator): Referral to a cardiac rehabilitation program outside of the safety net hospital setting.
  Interventions: Behavioral: Referral to an external cardiac rehabilitation program

INTERVENTIONS:
Behavioral: Tailored cardiac rehabilitation — The program will address the core components of CR.21 Each of the program components will have an individualized assessment with plan and goals set at the program intake visit. The 12-week program will alternate between group and individual sessions each week. Individualized plans will be reviewed every two weeks at the participant individual sessions. Group sessions will address physical activity, nutrition, and other program topics. Duration of the program was chosen to resemble a typical 12-week cardiac rehabilitation intervention. However, the program will have a greater emphasis on cultural tailoring, language concordance, lowering burden of real-time in-person attendance, motivational coaching, and addressing psychosocial needs.
  Arms: Tailored cardiac rehabilitation in a safety net setting
Behavioral: Referral to an external cardiac rehabilitation program — Participants will be referred to an external cardiac rehabilitation program outside of the safety net setting. This is the current standard of care.
  Arms: Referral to an outside cardiac rehabilitation program

SUMMARY:
The goal of this study is to determine whether participation in a tailored cardiac rehabilitation program delivered in a safety net setting, compared to usual care referral to an outside cardiac rehabilitation program, results in greater participation in cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+
2. Referred for cardiac rehabilitation for a covered indication:

   1. Acute myocardial infarction
   2. Percutaneous coronary intervention
   3. Coronary artery bypass surgery
   4. Heart valve repair or replacement
   5. Heart transplant
   6. Chronic stable angina
   7. Chronic systolic heart failure (EF <=35%)
3. Able to communicate in English, Spanish, or Cantonese
4. Able to consent for self

Exclusion Criteria:

1. Currently enrolled in hospice.
2. Provider says patient may not be approached for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Participation in at least 1 session of cardiac rehabilitation | 12 months
  In each arm, the proportion of participants who attended at least 1 cardiac rehabilitation session will be calculated.

SECONDARY OUTCOMES:
Completion of cardiac rehabilitation | 12 months
  In each arm, the proportion of participants who attend at least 2/3 of expected sessions of cardiac rehabilitation (24 sessions in the active comparator arm and 8 sessions in the experimental arm) will be calculated.
Change in six-minute walk distance | 12 months
  Change in distance walked in 6 minutes, following a standard protocol, from baseline to 12 months.
Change in six-minute walk distance | 3 months
  Change in distance walked in 6 minutes, following a standard protocol, from baseline to 3 months.
Change in quality of life | 12 months
  Change in PROMIS Global Health physical and mental subscores between baseline and 12 months. The PROMIS Global Health 10 questionnaire is a self-assessed questionnaire that asks participants to respond to 10 questions. The physical and mental health subscales each consist of four questions with a raw score between 4 and 20 that is converted to a standardized T-score. Higher scores represent better physical health.
Change in quality of life | 3 months
  Change in PROMIS Global Health physical and mental subscores between baseline and 3 months. The PROMIS Global Health 10 questionnaire is a self-assessed questionnaire that asks participants to respond to 10 questions. The physical and mental health subscales each consist of four questions with a raw score between 4 and 20 that is converted to a standardized T-score. Higher scores represent better physical health.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Beatty, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
At the conclusion of the study, we will follow local procedures and laws regarding the sharing of individual participant data. Any data that are shared will be de-identified prior to sharing.